CLINICAL TRIAL: NCT04482920
Title: The Effects of Hormone Therapy on Renal Hemodynamic Function in Transgender Youth
Brief Title: Effect of Hormone Therapy on Renal Function
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 20-0572
Record Dates: First submitted 2020-06-26; First posted 2020-07-23 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Transgenderism; Kidney Diseases; Kidney Injury
MeSH Terms: conditions — Transsexualism; Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transgender males: Transgender males who are clinically ready to start testosterone
  Interventions: Diagnostic Test: p-aminohippurate clearance study; Diagnostic Test: Iohexol infusion
- Transgender females: Transgender females who are clinically ready to start estradiol
  Interventions: Diagnostic Test: p-aminohippurate clearance study; Diagnostic Test: Iohexol infusion

INTERVENTIONS:
Diagnostic Test: p-aminohippurate clearance study — To measure kidney blood flow, small doses of a substance called p-aminohippurate (PAH) are used.
Diagnostic Test: Iohexol infusion — To measure glomerular filtration rate (GFR)

SUMMARY:
The purpose of this study is to understand the effects of testosterone or estradiol on kidney function in transgender adolescents and young adults.

ELIGIBILITY:
Inclusion Criteria:

* Identify as transgender
* Age 17-30 years (inclusive)
* Plan to start gender affirming hormone therapy (testosterone or estradiol) clinically in ≤ 1 months and remain on for at least 3 months

Exclusion Criteria:

* Cognitive, psychiatric or physical impairment resulting in inability to tolerate the study procedures (e.g. intellectual disability, schizophrenia, hallucinations)
* Type 1 or Type 2 diabetes
* Chronic kidney disease, or eGFR <60ml/min/1.73m2 by CKD-EPI formulation
* Uncontrolled hypertension (resting BP ≥ 140/90 mm/Hg)
* Allergy to shellfish, iodine or iohexol
* Currently taking: sulfonamides, procaine, thiazolesulfone and probenecid (renal clearance measurements of PAH cannot be made accurately if individuals are on these medications)
* Prior gender affirming hormone therapy use
* Prior gonadectomy
* Pregnancy

Ages: 17 Years to 30 Years | Sex: All
Age Groups: Child, Adult
Study Population: 20 transgender youth and young adults (10 transgender females, 10 transgender males) before and 3 months after initiation of gender affirming hormone therapy to determine the impact of gender affirming hormone therapy on intrarenal hemodynamic function and tubular function.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Change in measured glomerular filtration rate (GFR) | Baseline, 3 months

SECONDARY OUTCOMES:
Change in effective renal plasma flow | Baseline, 3 months
Change in biomarkers of tubular injury and repair (Neutrophil gelatinase-associated lipocalin [NGAL], Kidney injury molecule-1 [KIM-1], Chitinase-3-like protein 1 [YKL-40]) | Baseline, 3 months
Change in fat mass | Baseline, 3 months
  Quantified noninvasively by ImpediMed SFB7 single channel, tetra polar bioimpedance spectroscopy
Change in fat-free mass | Baseline, 3 months
  Quantified noninvasively by ImpediMed SFB7 single channel, tetra polar bioimpedance spectroscopy
Change in intracellular fluid | Baseline, 3 months
  Quantified noninvasively by ImpediMed SFB7 single channel, tetra polar bioimpedance spectroscopy
Change in extracellular fluid | Baseline, 3 months
  Quantified noninvasively by ImpediMed SFB7 single channel, tetra polar bioimpedance spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Natalie J Nokoff, MD, MSCS, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van Eeghen SA, Pyle L, Narongkiatikhun P, Choi YJ, Obeid W, Parikh CR, Vosters TG, van Valkengoed IG, Krebber MM, Touw DJ, den Heijer M, Bjornstad P, van Raalte DH, Nokoff NJ. Unveiling mechanisms underlying kidney function changes during sex hormone therapy. J Clin Invest. 2025 Mar 25;135(9):e190850. doi: 10.1172/JCI190850. eCollection 2025 May 1. PMID 40193283